CLINICAL TRIAL: NCT00168909
Title: Influence of Alfacalcidol on Falls in Elderly Postmenopausal, Alendronate-Treated, Osteopenic/Osteoporotic Women With High Risk of Falls
Brief Title: Influence of Alfacalcidol on Falls in Osteopenic/Osteoporotic Postmenopausal Women (ALFA Study)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Charite University, Berlin, Germany (Other)
Responsible Party: Prof. Dr. Dieter Felsenberg, Charité - Campus Benjamin Franklin, Centre for Muscle and Bone Research, Hindenburgdamm 30, 12200 Berlin, Germany
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ek.213-07 (IRB)
Record Dates: First submitted 2005-09-09; First posted 2005-09-15 (Estimated); Last update posted 2008-05-09 (Estimated); Status verified 2008-05

CONDITIONS: Osteoporosis, Postmenopausal; Osteopenia; Falls
Keywords: osteoporosis; frailty; falls
MeSH Terms: conditions — Osteoporosis, Postmenopausal; Bone Diseases, Metabolic; Osteoporosis; Frailty | interventions — alfacalcidol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): alfacalcidol 1µg/d
  Interventions: Drug: alfacalcidol
- 2 (Placebo Comparator): placebo
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: alfacalcidol — alfacalcidol 1 µg once daily, oral, for 3 years
  Arms: 1
Drug: placebo — placebo once daily, oral, for 3 years
  Arms: 2

SUMMARY:
The purpose of this study is to evaluate the effect of alfacalcidol 1 µg daily on the number of fallers in postmenopausal, alendronate-treated, osteopenic or osteoporotic women.

primary outcome = number of fallers (patients with at least one locomotor fall incl.mixed falls)

ELIGIBILITY:
Inclusion Criteria:

* age > 65 years
* postmenopausal women
* osteopenia/osteoporosis as defined by WHO criteria

Exclusion Criteria:

* Neoplasm or other severe diseases with life expectancy less than one year or expectation of rapid worsening within one year
* Chronic inflammatory rheumatoid disease
* Arthritis with continuous pain and influence on locomotion
* Inflammatory or metabolic bone disease, excluding osteoporosis.
* Subjects with antiosteoporotic medications who are not willing to switch over to alendronate treatment. Estrogen treatment can be continued
* 25-OH-Vitamin D3 < 12 ng/ml (12 ng/ml = 30 mmol/L)
* Systemic corticosteroid treatments of more than one month within previous 12 months
* Intolerability for alfacalcidol
* Hypercalcaemia (>2,7 mmol/l)
* Milk alkali syndrome
* Uncorrected, severe visual impairments
* Creatinin > 2.5 mg/dl (>220 µmol/L)

Min Age: 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 282 (Actual)
Dates: Start 2003-06; Primary Completion 2007-07 (Actual); Study Completion 2008-05 (Actual)

PRIMARY OUTCOMES:
primary outcome: number of fallers (patients with at least one locomotor fall incl.mixed falls) | 3 years

SECONDARY OUTCOMES:
secondary outcome: number of falls (locomotor falls, incl.mixed falls), all falls/fallers, neuromuscular parameters, BMD, biochemical parameters of calcium and bone metabolism; cognition and moods; muscle biopsies | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Dieter Felsenberg, Prof. Dr., Study Chair — Centre for Muscle and Bone Research, Charité - Campus Benjamin Franklin, Berlin, Germany
Locations (2):
- Germany (2):
  - Centre for Muscle and Bone Research, Charité - Campus Benjamin Franklin, Berlin
  - Centre for Muscle and Bone Research, Aerpah-Kliniken Esslingen, Stuttgart